CLINICAL TRIAL: NCT03184974
Title: Individualized Open Lung PEEP in Thoracic Surgery: A Prospective Multicenter Observational Study in 17 Spanish Hospitals
Brief Title: Open Lung PEEP in Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Carlos Ferrando, Principal investigador, Fundación para la Investigación del Hospital Clínico de Valencia
Other Study IDs: PEEPOPTIMA
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Thoracic Surgery; Ventilation Therapy; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During thoracic surgical procedures, while ventilating with a protective tidal volume, an open lung approach consisting of a recruitment maneuver followed by an individualized positive end-expiratory pressure (PEEP) titrated to best respiratory system compliance (Open-lung PEEP, OL-PEEP) would decrease driving pressure. To test this hypothesis, we performed a multicenter observational study in 17 Spanish teaching hospitals of patients undergoing one lung ventilation (OLV). In addition, we analyzed the association between the driving pressure and the prevalence of postoperative pulmonary complications (PPCs), and finally the association between the individualized PEEP and relevant patient preoperative or intraoperative variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing one lung ventilation

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing one lung ventilation during thoracic surgical procedures
Sampling Method: Probability Sample
Enrollment: 690 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | Postoperative. One week
  Atelectasis, acute respiratory failure, ARDS, pneumonia, reintubation, empyema, bronchospasm, pneumothorax, pneumonitis, bronchopleural fistula

SECONDARY OUTCOMES:
Descriptive analysis of the open lung PEEP | intraoperative
  Open lung PEEP is the PEEP of best dynamic respiratory system compliance during a PEEP titration trial

IPD SHARING:
Plan to Share IPD: Undecided